CLINICAL TRIAL: NCT05885854
Title: Exploratory Application of XTR003 as a Novel PET Myocardial Fatty Acid Metabolism Imaging Agent for the Detection of Viable Myocardium
Brief Title: XTR003 PET Radiotracer for the Detection of Viable Myocardium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sinotau Pharmaceutical Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STB-XTR003-201
Record Dates: First submitted 2022-12-25; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Ischemic Heart Disease (IHD)
Keywords: Coronary Artery Disease (CAD); Positron Emission Tomography (PET); XTR003 PET myocardial fatty-acid tracer; 18F-Fluorodeoxyglucose (18F-FDG); Non-ST-Segment Elevation Myocardial Infarction (NSTEMI); Old Myocardial Infarction (OMI); Total Coronary Occlusions (TCO)
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XTR003; At rest (Experimental): 1. Injection with XTR003 to investigate myocardial fatty-acid metabolism in patients with known IHD.
  2. Adjunct injection with 18F-FDG to investigate and trace myocardial glucose metabolism in patients with known IHD.
  The study population consisted of 50 participants from the following category of patients: (1) Patients with Non-ST elevation myocardial infarction (NSTEMI) (2) Patients with old myocardial infarction (3) Patients with total occlusions of coronary arteries.
  Interventions: Drug: XTR003

INTERVENTIONS:
Drug: XTR003 — Enrolled subjects were required to fast for ≥ 6 hours before drug administration at rest;
  1. Initial intravenous injection of 18F-FDG to each subject with a dose range of 2.0-3.0 mCi (74-111 MBq). Each patient will be imaged with PET for 10 minutes at 50-70 minutes after the injection.
  2. In few minutes, a single intravenous bolus injection of XTR003 will follow and administer to each patient with a dose range of 6.0-8.0 mCi (222-296 MBq). Each patient will be immediately imaged with PET for 15 minutes.

SUMMARY:
The study was designed to explore the clinical feasibility of XTR003, a PET myocardial fatty-acid tracer, for the detection of viable myocardium in patients with ischemic heart disease (IHD).

DETAILED DESCRIPTION:
The incidence of IHD is increasing in China and globally. However, the 18F-FDG-PET patient preparation protocols present challenges in certain patients such as patients with type I and II Diabetes Mellitus. XTR003 is a PET fatty-acid analog used in the imaging of myocardial fatty-acid metabolism. The combination of fasting XTR003/18F-FDG PET imaging may overcome the shortness of glucose-loaded 18F-FDG PET imaging protocol and effectively identify viable myocardium.

This is an exploratory, single-arm, open-label, phase II clinical study with the following objectives:

1. To explore the clinical feasibility of XTR003 for the detection of viable myocardium in patients with NSTEMI, old myocardial infarction, or total occlusions of coronary arteries.
2. To evaluate the safety and adverse events incidence of XTR003 in patients with known IHD.
3. To evaluate the sensitivity and specificity of fasting 18F-FDG/XTR003 PET combining imaging in detecting viable myocardium.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years old men and women.
2. The diagnosis and assessment of the disease meet any of the following criteria:

   (a) Patients who meet the diagnostic criteria for NSTEMI are stable and require further imaging. (b) Patients with old myocardial infarction confirmed by medical history or imaging examination and now in the stable stage. (c) Patients diagnosed with total coronary occlusions based on coronary angiography showing anterior flow occlusion segment with TIMI grade 0 or coronary CTA examination showing complete coronary artery occlusion.
3. The rest 99mTc-Sestamibi (MIBI) SPECT imaging has been completed in the past month and no imaging technical issues were leading to poor image quality. Image indicated myocardial perfusion defect of ≥ 2 segments or total resting perfusion score (SRS) ≥4.
4. The patient has completed glucose-loaded 18F-FDG myocardial metabolic PET imaging in the last month and has not failed to diagnose because of poor image quality due to technical problems with the imaging, except for his own glucose regulation.
5. Patients who can communicate properly with the investigators, understand and follow the study requirements, voluntarily participate, and understand and sign the informed consent.

Exclusion Criteria:

1. Patients with other preexisting cardiovascular diseases including but not limited to dilated or hypertrophic cardiomyopathy, pericarditis, aortic dissection, uncontrolled severe arrhythmias, and congenital heart disease are deemed not eligible for the study by the principal investigator.
2. Patients with severe acute or chronic lung disease, including but not limited to chronic obstructive pulmonary disease, asthma, bronchiectasis, emphysema, pulmonary fibrosis, pulmonary embolism, pneumonia, etc., are deemed not eligible for the study by the principal investigator.
3. Patients with severe or unstable central nervous system diseases, including but not limited to unstable cerebrovascular diseases, active epilepsy, infectious diseases of the central nervous system, and central nervous system, and central nervous system disease associated with neuropathy or limb movement disorders are deemed not eligible for the study by the principal investigator.
4. Patients with severe hemorrhagic diseases or coagulation disorders, including but not limited to purpura, hemophilia, and deficiency in vitamin K are deemed not eligible for the study by the principal investigator.
5. Patients with fever or active infectious diseases are deemed not eligible for the study by the principal investigator.
6. Patients with serious disorders of organ systems other than those described above and who are deemed not eligible for the study by the principal investigator.
7. Hematologic antigen/antibody test meets either of the following criteria: anti- HIV antibody (+) and syphilis antibody (+) are deemed not eligible for the study by the principal investigator.
8. Significant occupational exposure to or treatment with ionizing radiation (e.g., more than 50 mSv/yr) within 10 years.
9. Pregnant or lactating women.
10. People with mental disorders or poor compliance.
11. Men and women of reproductive age refused to adopt contraceptive plans during the study period and for 6 months after the study ended.
12. Other circumstances that the investigator considers inappropriate for participating in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2023-03-04 (Actual); Study Completion 2023-03-05 (Actual)

PRIMARY OUTCOMES:
To investigate the sensitivity of combining XTR003/FDG PET imaging | Day 1
  To simultaneously trace fatty-acid and glucose metabolisms for the detection of viable myocardium in IHD patients with NSTEMI, old myocardial infarction, or total occlusions of coronary arteries.
To investigate the specificity of combining XTR003/FDG PET imaging | Day 1
  To simultaneously trace fatty-acid and glucose metabolisms for the detection of viable myocardium in IHD patients with NSTEMI, old myocardial infarction, or total occlusions of coronary arteries.

SECONDARY OUTCOMES:
Number of study participants with treatment-related adverse events as determined by safety parameter changes according to CTCAE v5.0 | Up to 9 days
  Safety parameters included adverse events, vital signs (body temperature, blood pressure, respiration rate, pulse rate), physical examinations, laboratory tests (serum cardiac biomarkers, cardiac troponin I, serum biochemistry, haematology, and urinalysis) and electrocardiograms.

CONTACTS AND LOCATIONS:
Locations (1):
- TEDA International Cardiovascular Hospital, Tianjin, Tianjin Municipality, China